CLINICAL TRIAL: NCT05216471
Title: Diagnostic Accuracy of Chest X-ray in Coronavirus Disease 2019
Brief Title: Identify Coronavirus Disease by Chest X-ray
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelwahab Elsadek Ibrahim, Resident doctor, Assiut University
Other Study IDs: x-ray in covid19
Record Dates: First submitted 2022-01-27; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19 | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild illness: individuals who have any of the various signs and symptoms of covid-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and smell) but who do not have shortness of breath, dyspnea, or abnormal chest imaging findings .
  Interventions: Radiation: chest X-ray
- Moderate illness: individuals who show evidence of lower respiratory tract disease during clinical assessment or imaging and who have an oxygen saturation (SpO2) ≥94% on room air .
  Interventions: Radiation: chest X-ray
- Severe illness: individuals who have spO2<94% on room air, a ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2)<300 mm hg, respiratory frequency>30 breaths/min, or lung infiltrate >50%.
  Interventions: Radiation: chest X-ray

INTERVENTIONS:
Radiation: chest X-ray — Chest Xray : postero-anterior view ,digital high resolution X-ray or ,full inspiratory

SUMMARY:
to identify the diagnostic accuracy of chest X-ray in diagnosis of Coronavirus disease19 .

DETAILED DESCRIPTION:
The pandemic related to the coronavirus is now considered one of the deadliest epidemics. The numbers of cases exponentially increased with no specific treatment, creating havoc for the health and financial systems of the world [1-6]. Wuhan, the capital city of Hubei in China, reported the earliest cases that were treated as an unusual pneumonia. With the disease progression, the World Health Organization (WHO) announced the presence of several similar cases [7, 8]. Researchers revealed that a novel strain of the family Coronaviridae is the pathogen responsible for the respiratory illness of this disease and this is simulating two previous epidemics, namely MERS (Middle Eastern respiratory syndrome) and SARS (severe acute respiratory syndrome). The disease induced by SARS-CoV-2 was labelled as COVID-19 by the International Classification of Diseases (ICD) [9]. Chest radiographs are usually of limited value in the diagnosis of early stages especially in mild disease course; however, the CT findings may be present early even before the onset of the symptoms. Chest radiographs is very helpful in the intermediate to advanced stages of COVID-19 with features of acute respiratory distress syndrome (ARDS) as well as the follow-up [10-11]. This study to determine the COVID-19 disease course and severity using chest X-ray (CXR) scoring system and correlate these with patients' age, sex, and outcome.

ELIGIBILITY:
Inclusion Criteria:

* All individuals attending the Radiodiagnosis Department , who had paired posterior-anterior chest radiographs and RT-PCR nasopharyngeal swabs for COVID-19 at the time of initial attendance with moderate to advanced stage.
* The patients have positive finding in the posterior-anterior chest radiographs , multislice computer tomography and RT-PCR nasopharyngeal swabs for COVID-19.
* The patients with positive finding in the laboratory investigation (CBC, CRP ,ESR , S.Ferritin & D-Dimmer) .
* Patients with positive chest-CT finding and laboratory finding despite of having negative PCR swab

Exclusion Criteria:

* Patients exceeding 30 days after positive RT-PCR .
* Patients diagnosed with mediastinal lymphadenopathy , masses ,Tree in bud appearance ,Pneumothorax. Or Cavitation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will include 150 patients with suspected COVID-19 infection with positive RT_PCR, MSCT Chest , laboratory investigation. This sample size would be statistically significant. Each group comprises 50 patient , the radiolographic finding xray will be revising and tabulated in each one of the three group according to a standard scheme.
  the finding will be correlated with clinical and laboratory finding . statistic of collected data will be performed as needed .
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of initial CXR, where it is reported as having classic COVID-19 features in different clinical severity presentation correlation of xray finding with clinical and laboratory finding. | baseline
  to identify the accuracy of chest x-ray in diagnosis of classical covid19 according to the severity of the clinical presentation and laboratory finding

CONTACTS AND LOCATIONS:
Overall Officials: Nagham Nabil Mahmoud, Professor, Study Chair — Radiodiagnosis Department - Faculty of Medicine - Assiut University; Hosameldeen Abozaid Yousef, Associate Professor, Study Director — Radiodiagnosis Department - Faculty of Medicine - Assiut University; Aliaa Abd-Raboh Mohamed, Professor, Study Director — Department of Chest Diseases Faculty of Medicine - Assiut University; Mohamed abdelwahab Ibrahim, bachelor, Principal Investigator — Radiodiagnosis Resident, Assiut Chest Hospital
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
This sample size would be statistically significant. Each group comprises 50 patient , the radiolographic finding xray will be revising and tabulated in each one of the three group according to a standard scheme.
  the finding will be correlated with clinical and laboratory finding . statistic of collected data will be performed as needed .

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Custro N, Scafidi V, Borsellino T. [Changes in the thyroid hormone picture that may be found in severely decompensated type II diabetics]. Minerva Med. 1991 Jan-Feb;82(1-2):9-14. Italian. PMID 2000180
- [Background] Litmanovich DE, Chung M, Kirkbride RR, Kicska G, Kanne JP. Review of Chest Radiograph Findings of COVID-19 Pneumonia and Suggested Reporting Language. J Thorac Imaging. 2020 Nov 1;35(6):354-360. doi: 10.1097/RTI.0000000000000541. PMID 32520846
- [Background] Cheng VC, Lau SK, Woo PC, Yuen KY. Severe acute respiratory syndrome coronavirus as an agent of emerging and reemerging infection. Clin Microbiol Rev. 2007 Oct;20(4):660-94. doi: 10.1128/CMR.00023-07. PMID 17934078
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570